CLINICAL TRIAL: NCT06264934
Title: An Investigation Into Dielectric Assessment of Permittivity and Cancer in Human Using a Novel Electrical Capacitance Tomography Scanner
Brief Title: An Investigation Into Dielectric Assessment of Permittivity and Conductivity in Human Using a Novel Electrical Capacitance Tomography Scanner
Acronym: DiCECT
Status: Recruiting | Type: Observational
Sponsor: Zedsen Limited (Industry)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DiCECT
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Benign Breast Disease
Keywords: Breast Cancer; Electrical Capacitance Tomography; Permittivity
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part A: Twenty healthy participants will be recruited to examine the ability of the Z-scanner to identify healthy breast tissue and assess repeatability and reproducibility of the device.
  Interventions: Device: Breast scan using the Z-scanner
- Part B: 70 participants (35 benign and 35 malignant) will be recruited to investigate the ability of the Z-scanner to correctly identify and differentiate malignant and/or benign lesions from healthy breast tissue.
  Interventions: Device: Breast scan using the Z-scanner

INTERVENTIONS:
Device: Breast scan using the Z-scanner — Four repeated scans of both breasts using the Z-scanner.
  Groups: Part A
Device: Breast scan using the Z-scanner — A scan of both breasts using the Z-scanner.
  Groups: Part B

SUMMARY:
The goal of this observational study is to investigate the ability of a the Z-scanner to identify and differentiate cancer and benign lesions from healthy breast tissue based on permittivity. The main questions it aims to answer are:

1. Determine the permittivity values of the Z-scanner associated with healthy, benign, and malignant tissue in human breasts.
2. Determine the repeatability, reproducibility, inter-and intra-operator variability of the Z-scanner.

DETAILED DESCRIPTION:
Permittivity is the measure of a material's ability to store electrical energy in the electric field. Different materials are known to have different permittivity including the human body. Research is looking into utilising permittivity differences in the human body to detect cancer. There is a particular focus in breast cancer because it is the most common type of cancer in women globally, and research has shown that permittivity of healthy breast tissue is different to cancer tissue. Furthermore, breast tissue can be easily accessible by non-invasive means and has well-established tools available to support cancer detection. However, results from many studies vary greatly and more research is needed to understand how permittivity can be used in cancer research. Zedsen Limited has developed a permittivity measuring device (Z-scanner) capable of measuring a material's permittivity. The purpose of this study is to establish the permittivity of healthy, benign, and cancer tissue associated with the Z-scanner.

90 women attending a routine screening assessment clinic or a one stop clinic at Charing Cross Hospital will be recruited over the course of a year. The study is split into 2 parts. Part A will recruit 20 participants to assess whether scanner results can be repeated and reproduced by different users and hardware. Part B will recruit 70 participants to assess whether the Z-scanner can differentiate between benign and cancerous lesion. All participants will have both their breasts scanned using the Z-scanner during their routine appointment. This allows us to investigate the ability of the Z-scanner to identify and differentiate benign and cancerous lesions from healthy breast tissue based on permittivity. Results from this study can further our understanding on how permittivity and such devices can be used in cancer research.

ELIGIBILITY:
Inclusion Criteria:

* Attending a symptomatic clinic or other appointment at a participating breast clinic site
* Assigned female sex at time of birth
* Aged 18 years or older at time of scan
* Willing, able and mentally competent to read, understand, and provided informed consent in English

Exclusion Criteria:

* Participants who have undergone biopsy less than 14 days before the Z-scanner scan
* Participants with implanted electronics
* Participants with breast implants
* Participants with nipple piercings (unless they are removed prior to the scan)
* Participants who are lactating
* Pregnant participants by verbal confirmation
* Participants with pacemakers
* Participants with open breast wound
* Participants who had previous breast surgery (mastectomy, lumpectomy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 healthy participants 35 participants with benign lesions 35 participants with malignant lesions
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of complex permittivity of breast tissue components | Jan-Nov 2024
  Permittivity will be estimated from a series of inter-electrode capacitance derived from raw outputs of the Z-scanner using in house algorithms.

SECONDARY OUTCOMES:
Permittivity target-to-background contrast ratios for targets of interest (e.g. malignant lesion, benign lesion) | Jan-Nov 2024

OTHER OUTCOMES:
Repeatability of the Z-scanner | Jan-Nov 2024
  Response voltage signals from raw output of the Z-scanner will be compared between each repeated breast scans.
Reproducibility of the Z-scanner | Jan-Nov 2024
  Response voltage signals from raw output of the Z-scanner will be compared between breast scans obtained by different Z-scanners and different operators.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No